CLINICAL TRIAL: NCT01498406
Title: Vitamin D Status, Disease Specific and Quality of Life Outcomes in Patients With Cutaneous Lupus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: secondary to funding issues and low enrollment
Sponsor: Emory University (Other)
Collaborators: Dermatology Foundation (Other)
Responsible Party: Principal Investigator, Laura K. DeLong, MD, MPH, Assitant Professor of Dermatology, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00051622
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-06

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: cutaneous lupus erythematosus; vitamin D; quality of life
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high dose vitamin D3 (Experimental): 4,000 IU of vitamin D3 daily for 8 months
  Interventions: Dietary Supplement: vitamin D
- low dose vitamin D3 (Active Comparator): 400 IU of vitamin D3
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — The investigators will carry out a two-armed prospective pilot study of the influence of vitD on cutaneous lupus (CLE) disease severity. Patients with CLE will be eligible for an observational or interventional arm based on their 25(OH)D levels and consent. Subjects with low vitD status (<30 ng/mL) will be eligible for the investigational arm involving participation in a randomized controlled trial of daily high dose (4000 IU) vs. low dose (400 IU) vitD supplementation for 8 months. Subjects who have sufficient vitD status (>30ng/mL) or those with low vitD who choose not to participate in the RCT are eligible for continued participation in the observational arm of the study. All subjects will be followed at 4, 8, and 12 months.
  Other Names: The investigators will be using vitamin D soft gels in 400 IU and 4,000 IU provided by Carlson laboratories.

SUMMARY:
Lupus is a disease in which the immune system, which normally fights infection, begins to attack healthy cells in the body. This phenomenon is called autoimmunity and what the immune system attacks is called the autoantigen. Lupus can affect many parts of the body and often affects the skin, with immune cells attacking autoantigens in the skin and causing a rash. This rash is often visible to the public because it tends to occur on sun-exposed areas, for example a patient's face, chest, and arms. For this reason, among others, skin lupus can be a source of disability and poor health related quality of life in many patients with this disease. It is not completely understood why or how someone might develop lupus, however there are likely many reasons which include their genetics and also the kind of environment they live in.

One such environmental factor, vitamin D, is more commonly known as a vitamin important for bone health. However, we are learning that vitamin D has effects all over the body, and is also important for a healthy immune system. Low levels of vitamin D have been associated with an increased risk of other autoimmune disorders such as diabetes and multiple sclerosis, and have also been found to be common in skin lupus patients.

Vitamin D is made in the skin when it is exposed to the sun, specifically ultraviolet B radiation (UVB). The main source of vitamin D for most people is its production in the skin because the normal American diet is not high in vitamin D. However, patients with skin lupus tend to stay out of the sun because their rash is made worse by sunlight, which is thought to produce more of the autoantigens in the skin attacked by the immune system. Additionally, as skin doctors (dermatologists) we recommend sun protection to skin lupus patients to minimize sun-sensitivity and prevent flares of their skin disease. However we may be putting them at risk for low vitamin D status and even more severe disease. Another risk factor that puts skin lupus patients at risk for vitamin D deficiency is that these patients generally have darker skin types which blocks UVB and further limits vitamin D production in the skin.

Given that skin lupus patients are at high risk for low vitamin D status as mentioned above, the investigators propose a research study that will provide information about vitamin D levels in these patients. The investigators seek to identify how many skin lupus patients have low vitamin D status and how vitamin D influences the natural history of this skin disease. Additionally the investigators will evaluate whether or not supplementation with high dose vitamin D will lessen the severity and negative quality of life impact of skin lupus. Supplementation of vitamin D by mouth is an inexpensive, well tolerated, and safe over the counter method to replete and maintain a normal vitamin D status. Studies in other autoimmune diseases, specifically Crohn's disease and multiple sclerosis, have shown that high dose vitamin D supplementation improves disease severity. It is the hope of the investigators that this will also be observed in skin lupus patients.

In summary, the investigators seek to move beyond establishing an association between vitamin D status and skin lupus. The investigators aim to elucidate the therapeutic benefit, if any, of vitamin D status on disease severity and quality of life while controlling for important factors that may influence vitamin D status. If the investigators are to show improvement in disease severity with vitamin D supplementation, this would be a cost-effective additional therapy to our standard clinical practice. Future research would also allow us to investigate other alternative markers of vitamin D deficiency and disease activity in skin lupus patients, a population at high risk for low vitamin D status and in need of further research.

ELIGIBILITY:
i. Inclusion Criteria for observational arm:

* Sites: Subjects will be primarily recruited from the Emory and Grady Memorial Hospital Dermatology Clinics. Additional recruitment will be from community dermatologists using a flyer since this is a relatively uncommon skin disease. This study will also be listed on the NIH and Lupus Foundation of America websites.
* Stage of Disease: A previous or new diagnosis of CLE, either clinically supported or confirmed by skin biopsy.
* Age: Adult subjects, greater than 18 years old.

ii. Inclusion criteria for control group in observational arm: Dermatology patients with skin disease, but without CLE, with skin types IV, V, VI will be recruited for the control group.

iii. Inclusion criteria for interventional arm: Patients with 25(OH)D levels <30ng/ml.

iv. Exclusion Criteria:

* Patients who are already actively having their vitD levels monitored and repleted.
* Patients with 25(OH)D levels ≥30 ng/ml will be excluded from the RCT but are eligible for the observational arm of the study.
* Patients with systemic lupus as defined by the American Rheumatism Association criteria.
* Patients with renal lithiasis, hypercalcemia, inflammatory bowel disease, or sarcoidosis.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
cutaneous lupus severity as measured by the CLASI instrument(Cutaneous Lupus Erythematosus Disease Area and Severity Index) | 1 year
  The CLASI (Cutaneous Lupus Erythematosus Disease Area and Severity Index) is a validated CLE disease severity measure that has been in use in clinical trials since 2005. This scale captures cutaneous, mucosal membrane, and alopetic disease activity (erythema and scale/hypertrophy) as well as damage (dyspigmentation and scarring/ atrophy/ panniculitis).

SECONDARY OUTCOMES:
Quality of life as measured by the Skindex 29 | 1 year
  No cutaneous lupus specific quality of life (QOL) measure exists, but the Skindex 29, a validated skin-specific QOL measure has been used in previous studies along with three added questions: two related to patient concerns about photosensitivity and one related to patient concerns about hair loss. The investigators propose to use the Skindex-29, with three independent scores that can be used in the measurement of health related QOL in dermatological patients.
serum 25-hydroxy vitamin D | 1 year
  a blood test to asses 25-hydroxy vitamin D level

CONTACTS AND LOCATIONS:
Overall Officials: Laura K DeLong, MD, MPH, Principal Investigator — Emory Dermatology
Locations (1):
- Emory Dermatology Clinics, Atlanta, Georgia, United States